CLINICAL TRIAL: NCT02202304
Title: The Effects of Chlorhexidine/Thymol Varnish on the Abutment Teeth in Partial Denture Wearers.
Brief Title: The Effects of Chlorhexidine/Thymol Varnish on Partial Denture Patient
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Researcher changed jobs. Unable to carry out the project
Sponsor: Rosa Moreno Lopez (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor-Investigator, Rosa Moreno Lopez, Dr, University of Aberdeen
Organization: University of Aberdeen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHLOVADENT
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Periodontal Disease; Caries
MeSH Terms: conditions — Periodontal Diseases | interventions — Chlorhexidine; chlorhexidine, thymol drug combination; Thymol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine/Thymol varnish (Experimental): Participants to the study will receive an application of either the placebo or the product being studied every 3 months. This will be applied on all abutment teeth using a microbrush by "painting" it over the surfaces of these teeth.
  Interventions: Drug: Chlorhexidine/Thymol varnish
- Placebo varnish (Placebo Comparator): Participants to the study will receive an application of either the placebo or the product being studied every 3 months. This will be applied on all abutment teeth using a microbrush and "painting" it on all the surfaces of these teeth..
  Interventions: Drug: Chlorhexidine/Thymol varnish

INTERVENTIONS:
Drug: Chlorhexidine/Thymol varnish — This will be applied on abutment teeth on partial denture wearers every 3 months during a period of 2 years.
  Other Names: Cervitec Plus (1% chlorhexidine plus 1% thymol)

SUMMARY:
Cervitec, a chlorhexidine based varnished has been proven to reduce caries risk in younger populations. This study wants to investigate if the use of this product would reduce the risk of losing abutment teeth on patients that are wearing partial dentures as the literature has proven that these teeth are more prone to caries and periodontal disease.

The primary objectives of this research project are to:

1. Assess if the topical application of CHX/thymol varnish every three months on partial denture abutment teeth results in a clinicallu significant decrease in any loss of attachment compared to no application, and
2. Assess if the topical application of CHX/thymol vanirhs every three months on partial denture abutment teeth results in a clinically significant decrease in carious lesion development or progression compared to no application.

The secondary objectives of this research project are to:

1. Assess of the topical application of CHX/thymol varnish every three months on partial denture abutment teeth compared to no application results in a clinically significant difference in:

1. Bleeding on probing (BoP).
2. Plaque formation.
3. Periodontal pocket depths.
4. Microbial composition and GCF cytokine profile of the sub gingival environment.
5. The patients self perception of oral health.

DETAILED DESCRIPTION:
* 2 baseline samples of the Gingival Crevicular Fluid (GCF) and the subgingival samples. The first baseline sample will be done on the day of the first impressions and the second one the day of denture fitting.
* The following information will be recorded on the CRFs: Silness and Löe Plaque index, BoP, probing depth, clinical attachment level, LoA, Kennedy classification, material of the partial denture and type of clasp (or no clasp) and ICDAS code.
* The patient will also fill in the OHIP-14 questionnaire (Oral Health Impact Profile) to assess their self perception of oral health.
* A photograph of the abutment teeth and the partial denture will be taken.
* We will also take a full history of the patient including: name, DOB and medications.
* The GCF and subgingival sampled will be taken every 6 months on the appointment where the varnish is applied.
* All the laboratory samples will be labelles with the same identification number that the patient has been allocated and a date will also be written on it. All the samples will be analysed in Plymouth and stored in a - 50°C freezer (the samples taken at the University of Aberdeen will be stored in the same type of freezer and shipped periodically to the Penninsula University for tests maintaining the same temperature conditions). They will be testing the microbial composition and GCF cytokine profile of the sub gingival environment
* All measurements will be reassessed at 12 months and 24 months. In addition to the denture hygiene index: Budtz-Jørgensen (1977) Index (plaque accumulation on the denture).

The data will be collected by one clinician in each dental school. All clinicians will be calibrated appropriately.

Calibration: Before any examination starts we will assess the consistency of each examiner (intra-exmainer) and also the variation between exmainers (inter-exmainer reproducibility). Each examiner will independently examiner the same group of 20 subjects and compare his or her findings. When findings contain major discrepancies, subjects should be recalled in order that differences in diagnoses can be reviewed by the exmainers and resolved by group discussion. If certain examiners consistently produce significantly different results from the majority, and attmepts to correct their performance fail, they will be excluded from the team. It will be made clear to all potential examiners, before these exmainations begin, that ability to standardize examination results is not a measure of clinical skills (Oral Health Surveys 4th edition. WHO. Geneva 1997) All the data will be recorded on the case report forms (CRFs).

ELIGIBILITY:
Inclusion Criteria:

* Patients that are going to have a new denture fitted at the Dental School of the University of Aberdeen and Penninsula Dental School.
* Patients aged 18 years or over.

Exclusion Criteria:

* Patients that already have a denture.
* Patients that are taking antibiotics.
* Patients allergic to any of the components of the products.
* Pregnant women.
* Severe systemic illness.
* Patient with active periodontal disease (BoP and pockets ≥3mm) on abutment teeth.
* Presence of caries on abutment teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-10 (Estimated); Primary Completion 2019-09-10 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Assess if the topical application of CHX/thymol varnish every three months on partial denture abutment teeth results in a clinicallu significant decrease in any loss of attachment compared to no application | Assesed at the begining, at 12 months and at 24 months
  we will measure the Loss of Attachment (LoA) around each abutment tooth at 6 points

SECONDARY OUTCOMES:
Assess if the topical application of CHX/thymol vanirhs every three months on partial denture abutment teeth results in a clinically significant decrease in carious lesion development or progression compared to no application | at the beginning, at 12 months and at 24 months
  We will record the presence of dental caries using ICDAS

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Moreno Lopez, BDS, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
within 6 months

REFERENCES:
- [Background] Baca P, Clavero J, Baca AP, Gonzalez-Rodriguez MP, Bravo M, Valderrama MJ. Effect of chlorhexidine-thymol varnish on root caries in a geriatric population: a randomized double-blind clinical trial. J Dent. 2009 Sep;37(9):679-85. doi: 10.1016/j.jdent.2009.05.001. Epub 2009 May 13. PMID 19497653
- [Background] Tanaka J, Tanaka M, Kawazoe T. Longitudinal research on the oral environment of elderly wearing fixed or removable prostheses. J Prosthodont Res. 2009 Apr;53(2):83-8. doi: 10.1016/j.jpor.2008.10.003. Epub 2009 Jan 10. PMID 19318078
- [Background] Shimura Y, Wadachi J, Nakamura T, Mizutani H, Igarashi Y. Influence of removable partial dentures on the formation of dental plaque on abutment teeth. J Prosthodont Res. 2010 Jan;54(1):29-35. doi: 10.1016/j.jpor.2009.08.003. Epub 2009 Oct 8. PMID 19818702
- [Background] Clavero J, Baca P, Paloma Gonzalez M, Valderrama MJ. Efficacy of chlorhexidine-thymol varnish (Cervitec) against plaque accumulation and gingival inflammation in a geriatric population. Gerodontology. 2006 Mar;23(1):43-7. doi: 10.1111/j.1741-2358.2006.00085.x. PMID 16433641